CLINICAL TRIAL: NCT02503085
Title: A Randomized, Single-dose, 4-way Crossover, Open-label, Pharmacokinetic (PK) Study Comparing a 2% (w/v) Suspension of Ibuprofen (400 mg/20 mL Nurofen for Children®) With a Swiss Reference 2% (w/v) Suspension of Ibuprofen (400 mg/20 mL Algifor Dolo Junior®) in the Fed and Fasted States
Brief Title: Ibuprofen Suspension Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL1304; 2013-003366-14 (EudraCT Number)
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteer Study
Keywords: Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nurofen for Children® (fasted) (Experimental): Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted condition
  Interventions: Drug: Nurofen for Children®
- Nurofen for Children® (fed) (Experimental): Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fed condition
  Interventions: Drug: Nurofen for Children®
- Algifor Dolo Junior® (fasted) (Active Comparator): Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted condition
  Interventions: Drug: Algifor Dolo Junior®
- Algifor Dolo Junior® (fed) (Active Comparator): Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fed condition
  Interventions: Drug: Algifor Dolo Junior®

INTERVENTIONS:
Drug: Nurofen for Children®
  Other Names: Ibuprofen orange oral suspension
  Arms: Nurofen for Children® (fasted); Nurofen for Children® (fed)
Drug: Algifor Dolo Junior®
  Other Names: Ibuprofen oral suspension
  Arms: Algifor Dolo Junior® (fasted); Algifor Dolo Junior® (fed)

SUMMARY:
The purpose of this study was to determine the rate and extent of absorption of Ibuprofen suspension formulations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have given written informed consent.
* Age: ≥18 years ≤50 years.
* Sex: Male or female subjects are eligible for entry.
* Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use an effective method of contraception,
* Female subject of non-child bearing potential with negative pregnancy test at the screening visit
* Male subject willing to use an effective method of contraception, unless anatomically sterile
* Status: Healthy subjects as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Healthy Subjects with a Body Mass Index (BMI) of ≥20 and ≤27 kg/m2

Exclusion Criteria:

* Pregnancy or lactating female subjects.
* A history of significant disease of any body system.
* Any condition that may currently interfere with the absorption, distribution, metabolism or excretion of drugs.
* A history of allergy or intolerance related to treatment with ibuprofen, aspirin or other Non-Steroidal Anti-inflammatory Drug,or the excipients of the formulations.
* A history of or active peptic or duodenal ulcers or gastro-intestinal bleed or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders.
* A history of frequent dyspepsia, e.g. heartburn or indigestion.
* A history of migraine.
* Current smokers and ex-smokers who have smoked within 6 months.
* A history of drug abuse (including alcohol).
* High consumption of stimulating drinks (caffeine intake per day above 300 mg).
* Those with positive drugs of abuse screen including alcohol on any occasion throughout the study.
* Ingestion of a prescribed drug at any time in the 14 days before dosing with study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers during the previous month (such as barbiturates, carbamazepine, erythromycin, phenytoin, etc.).
* Ingestion of an over-the-counter preparation within 7 days before dosing with study medication.
* Donation of blood in quantity in the previous 12 weeks before enrolment into the study.
* Known human immune deficiency virus (HIV) positive status, or a positive viral serology screen.
* Topical use of ibuprofen within 7 days before dosing with study medication.
* Those previously randomised into this study.
* Employee at study site.
* Partner or first degree relative of the Investigator.
* Those who have participated in a clinical trial in the previous 12 weeks.
* Those unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2015-08-25 (Actual); Study Completion 2015-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Reckit Benckiser, Hull, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 60 subjects were screened and among them 16 subjects were screen failure, 2 subjects withdrew consent and 14 subjects were reserve.
Groups:
- Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior®: B = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted condition.
  A = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fed condition.
  C = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fed condition.
  D = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted condition.
- Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior®: D = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted condition.
  C = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fed condition.
  A = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fed condition.
  B = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted condition.
- Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior®: C = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fed condition.
  B = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted condition.
  D = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted condition.
  A = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fed condition.
- Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®: A = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fed condition.
  D = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted condition.
  B = Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted condition.
  C = Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fed condition.
Period: Period 1
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 1: Washout (3 to 7 Days)
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2: Washout (3 to 7 Days)
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 7 | 7 | 7 | 7
Completed | 6 | 7 | 6 | 7
Not Completed | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Period: Period 3
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 6 | 7 | 6 | 7
Completed | 6 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3: Washout (3 to 7 Days)
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 6 | 7 | 6 | 7
Completed | 6 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1-BACD: Nurofen for Children® - Algifor Dolo Junior® | Sequence 2-DCAB: Nurofen for Children® - Algifor Dolo Junior® | Sequence 3-CBDA: Nurofen for Children® - Algifor Dolo Junior® | Sequence 4-ADBC: Nurofen for Children® - Algifor Dolo Junior®
Started | 6 | 7 | 6 | 7
Completed | 6 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted and fed conditions.
  Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted and fed conditions.
Arm/Group | Overall Study
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.46 (8.660)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 28
Weight [Mean (Standard Deviation); unit: kg] | 70.88 (10.909)
Height [Mean (Standard Deviation); unit: m] | 1.711 (0.1000)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 24.07 (1.884)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: Analysis population included only subjects with evaluable plasma concentrations per treatment and who had taken at least one dose of medication in each treatment groups.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted): Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fasted condition.
- Treatment A: Nurofen for Children® 400 mg/20 mL (Fed): Nurofen for Children® suspension 400 mg/20 mL single-oral dose under fed condition.
- Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted): Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fasted condition.
- Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed): Algifor Dolo Junior® suspension 400 mg/20 mL single-oral dose under fed condition.
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
ng/mL | 37499.938 (8983.3020) | 26207.273 (5788.1116) | 34752.646 (5205.5859) | 26377.382 (7496.1966)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Administration to the Last Quantifiable Concentration at Time t (AUC0-t)
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
min*ng/mL | 6139350.787 (1315534.5598) | 5783712.850 (1251017.0271) | 5912050.421 (1353655.3076) | 5639716.354 (1533625.9496)

3. Secondary Outcome: Elimination Rate Constant (Kel)
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/min
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
1/min | 0.00599 (0.001238) | 0.00533 (0.001142) | 0.00602 (0.001221) | 0.00557 (0.001156)

4. Secondary Outcome: AUC From Administration to Infinity (AUC0-inf)
Description: AUC0-inf = AUC0-t + (Ct/Kel), where Ct was the last quantifiable concentration at time t.
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min*ng/mL
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
min*ng/mL | 6215205.302 (1324821.9469) | 5927787.749 (1283566.5280) | 5986690.115 (1379614.0039) | 5733877.552 (1536788.1908)

5. Secondary Outcome: Ratio of AUC0-t/AUC0-inf (AUCR)
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
Ratio | 0.988 (0.0059) | 0.976 (0.0184) | 0.988 (0.0074) | 0.983 (0.0118)

6. Secondary Outcome: Time to Cmax (Tmax)
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
min | 46.4 (17.33) | 72.0 (33.70) | 52.3 (40.91) | 71.7 (48.72)

7. Secondary Outcome: Plasma Concentration Half-life (T1/2)
Description: Terminal elimination half-life (T1/2) = ln(2)/Kel
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
min | 121.122 (28.6677) | 137.555 (37.6325) | 120.879 (30.5194) | 130.460 (30.7138)

8. Secondary Outcome: Plasma Concentration at Each Planned Nominal Time-point (Cn)
Description: Cn was derived using linear interpolation from the 2 samples taken either side of the nominal time where there was a sampling time deviation. For concentrations that were missing due to blood samples not being taken Cn was not derived.
Time Frame: Pre-dose, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480, 720 and 1440 mins (Day 1, Post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
ng/mL
  Time Post-Dose - 10 min | 5934.077 (6885.8643) | 5473.173 (7955.4756) | 5579.436 (5074.7709) | 4647.090 (6289.5788)
  Time Post-Dose - 15 min | 12315.358 (10819.4956) | 8486.946 (9318.9385) | 12251.837 (9535.7628) | 8566.950 (8227.2989)
  Time Post-Dose - 20 min | 18776.528 (13893.1674) | 11491.148 (10579.5320) | 18346.910 (12216.1356) | 11489.917 (8402.4627)
  Time Post-Dose - 30 min | 27860.671 (12228.9507) | 16171.896 (10459.1021) | 27557.463 (10049.7928) | 17619.547 (10451.6496)
  Time Post-Dose - 40 min | 31484.356 (7963.3886) | 20109.864 (9451.0500) | 31258.579 (7630.5525) | 21794.588 (10810.9958)
  Time Post-Dose - 50 min | 32538.663 (9976.7494) | 22216.449 (8667.4972) | 31026.608 (6935.4647) | 23041.910 (10063.5154)
  Time Post-Dose - 60 min | 30424.660 (5407.6867) | 22645.898 (7482.6836) | 28751.529 (6440.3355) | 22226.638 (7893.6789)
  Time Post-Dose - 70 min | 28817.725 (4189.7125) | 22585.564 (6387.2660) | 26979.890 (6495.2967) | 21619.517 (6805.8715)
  Time Post-Dose - 80 min | 27236.542 (4944.7693) | 21532.327 (5367.9576) | 25528.950 (6286.8439) | 21132.032 (6103.8828)
  Time Post-Dose - 90 min | 26045.659 (4445.1832) | 20697.612 (4961.1992) | 24080.631 (6464.0707) | 20182.637 (5379.6131)
  Time Post-Dose - 105 min | 23391.182 (4298.8943) | 19525.222 (3347.9779) | 22336.377 (5049.6930) | 18500.837 (4736.1272)
  Time Post-Dose - 120 min | 20702.122 (4461.6587) | 18414.660 (3038.3137) | 20053.854 (4561.3611) | 17112.477 (4579.0063)
  Time Post-Dose - 180 min | 14091.791 (3856.4139) | 13597.701 (3653.1273) | 13062.561 (3345.8475) | 12893.527 (3436.8623)
  Time Post-Dose - 240 min | 9649.611 (2767.9584) | 10997.109 (3518.9434) | 9483.481 (3427.9947) | 9895.761 (3586.4589)
  Time Post-Dose - 360 min | 3992.230 (1611.5462) | 5390.090 (2071.2073) | 3830.211 (1667.1184) | 5612.610 (4105.1920)
  Time Post-Dose - 480 min | 1942.286 (948.4031) | 2839.215 (1352.4747) | 1930.929 (1069.7491) | 2650.093 (1697.3457)
  Time Post-Dose - 720 min | 560.199 (343.2360) | 829.589 (460.9511) | 544.660 (417.5077) | 788.223 (646.7288)
  Time Post-Dose - 1440 min | 127.547 (34.2600) | 149.707 (36.4129) | 189.103 (85.3662) | 145.298 (15.3467)

9. Secondary Outcome: Number of Subjects With Adverse Events (AEs).
Description: Intensity was determined by the Investigator. For symptomatic AEs the following definitions were applied.
  Mild = AE did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/pain.
  Relationship to Investigational Medicinal Products (IMP)
  Unassessable/Unclassified = Insufficient information to be able to make an assessment.
  Conditional/ Unclassified = Insufficient information to make an assessment at present.
  Unrelated = No possibility that AE was caused by IMP. Unlikely = Slight, but remote, chance that AE was caused by IMP. Possible = Reasonable suspicion that the AE was caused by IMP. Probable = Most likely that AE was caused by IMP. Certain = AE was definitely caused by IMP.
Time Frame: Up to follow-up day 7
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment B: Nurofen for Children® 400 mg/20 mL (Fasted) | Treatment A: Nurofen for Children® 400 mg/20 mL (Fed) | Treatment D: Algifor Dolo Junior® 400 mg/20 mL (Fasted) | Treatment C: Algifor Dolo Junior® 400 mg/20 mL (Fed)
Number analyzed (Participants) | 27 | 28 | 27 | 26
Participants
  Treatment Emergent Adverse Event (TEAE) | 3 | 4 | 7 | 3
  Serious TEAE | 0 | 0 | 0 | 0
  TEAE Leading to Withdrawal | 0 | 1 | 1 | 0
  Intensity - Mild | 3 | 2 | 6 | 2
  Intensity - Moderate | 0 | 2 | 0 | 1
  Intensity - Severe | 0 | 0 | 1 | 0
  Relationship to IMP - Certain | 0 | 0 | 0 | 0
  Relationship to IMP - Probable | 0 | 0 | 0 | 0
  Relationship to IMP - Possible | 0 | 1 | 0 | 1
  Relationship to IMP - Unlikely | 1 | 2 | 2 | 1
  Relationship to IMP - Unrelated | 2 | 1 | 5 | 1
  Relationship to IMP - Conditional/Unclassified | 0 | 0 | 0 | 0
  Relationship to IMP - Unassessable /Unclassifiable | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to follow-up day 7
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=28)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Feeling cold (General disorders) | 1 (1)
Peripheral swelling (Gastrointestinal disorders) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No